CLINICAL TRIAL: NCT05359588
Title: Association Between Postoperative Cerebral Vascular Complication and Functional Prognosis and Cerebral Small Vascular Disease (CSVD) After Thoracic Surgery : an Exploratory Study
Brief Title: Functional Prognosis of Post-operative Patients With Cerebral Small Vascular Disease(CSVD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSVD2021
Record Dates: First submitted 2022-01-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Small Vessel Diseases; Long Term Adverse Effects
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Long Term Adverse Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators perform a retro-prospective exploratory cohort study among patients 65 to 85 years old with pre-operative head MRI result after thoracic surgery in Renji Hospital Affiliated to Shanghai Jiaotong University from November 2020 to December 2021. Perioperative data were collected, including preoperative general condition, laboratory examination, auxiliary examination (blood routine, blood coagulation, liver and kidney function, etc.), perioperative indicators （use of anesthetics, anesthetic time, blood pressure, etc.）, postoperative cerebral function follow-up and occurrence of cerebral vascular complications (brain infarction, brain bleed, etc.) of patients.

ELIGIBILITY:
Inclusion Criteria:

* 65≤age<85
* after thoracic surgery
* finish pre-operative brain MRI

Exclusion Criteria:

* mental illness
* existing dementia and other diseases: Alzheimer disease, dementia, Parkinson's disease, Huntington's disease, systemic lupus erythematosus, etc.
* previous cerebral infarction or hemorrhage

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all postoperative patients between 65 and 85 years old with pre-operative brain MRI results in Renji Hospital Affiliated to Shanghai Jiaotong University from November 2020 to December 2021 after thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative overt stroke | 1 year after surgery
  Postoperative overt stroke detected by MRI of the brain

SECONDARY OUTCOMES:
Physical function after surgery as assessed using Activities of Daily Living (iADL) Scale | 1 year after surgery
  score of Activity of Daily Living Scale with total score of 78, higher score, better function) and Modified Ranking Scale from 0(no symptomatic post-infarction complication ) to 6 (death after cerebral infaction)
Physical function after surgery as assessed using the Modified Rankin Scale | 1 year after surgery
  The scale runs from 0-6, running from perfect health without symptoms to death. A higher score is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China